CLINICAL TRIAL: NCT02098577
Title: Effect of Two Different Rehabilitation Programs on Balance in Parkinsonian Patients: Crossover Versus Stabilometric Platform
Brief Title: Crossover Versus Stabilometric Platform in Parkinson's Disease
Acronym: PDvsCOPD
Status: Completed | Type: Observational
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor
Other Study IDs: PDvsCOPD; PDvsCOPD (Other: Ospedale generale di zona "Moriggia-Pelascini")
Record Dates: First submitted 2014-03-22; First posted 2014-03-28 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Parkinson's Disease
Keywords: Balance
MeSH Terms: conditions — Parkinson Disease | interventions — Crossing Over, Genetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PD patients cross-over treatment: 30 PD patients (according to Gelb et al) in Hoen&Yahr stage 3, underwent cross-over treatment with the ability to walk without any assistance with mini-mental state examination score >26.
  Interventions: Other: Crossover
- PD patients stabilometric platform: 30 PD patients (according to Gelb et al) in Hoen&Yahr stage 3, underwent stabilometric platform treatment, with the ability to walk without any assistance with mini-mental state examination score >26.
  Interventions: Other: Stabilometric Platform

INTERVENTIONS:
Other: Crossover — Crossover cycle
  Groups: PD patients cross-over treatment
Other: Stabilometric Platform — This Stabilometric plate allows to assess the balance with an objective and reliable measurement, in both standard static or dynamic unstable condition
  Groups: PD patients stabilometric platform

SUMMARY:
The aims of this study is to assess the efficacy of the crossover on balance in Parkinsonian patients and compare this results with the results of a control group of patients treated with a stabilometric platform.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disorder characterized by different motor symptoms (rigidity, akinesia, tremor and impairment of balance and gait). Even though pharmacological treatment has changed the natural course of the disease, balance worsens over time and leads to falls. The aims of this study is to assess the efficacy of the crossover (group 1) on balance in Parkinsonian patients and compare this results with the results of a control group of patients treated with a stabilometric platform (group 2). The group 1 executed 6 days/week for a 4-weeks cycle a crossover protocol based on the first 4 level of resistance and a training which lasts at most 5 minutes. The group 2 executed 6 days/week for a 4-weeks cycle different exercises with the stabilometric platform in monopodalic and in bipodalic standing.

ELIGIBILITY:
Inclusion Criteria:

* PD in stage III Hoen&Yahr according to Gelb et la. with the ability to walk without any assistance and with Mini Mental State Examination (MMSE) score > 26

Exclusion Criteria:

* MMSE < 26
* Coexistence of other neurological diseases
* PD patients with relevant orthopedic, rheumatic and muscular conditions

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients with PD in stage III Hoen&Yahr according to Gelb et la. with the ability to walk without any assistance and with Mini Mental State Examination (MMSE) score > 26.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
BBS | One month
  Berg Balance Scale

SECONDARY OUTCOMES:
6MWT | One month
  Six minutes walking test
TUG | One month
  Time up and Go test
UPDRS II | One month
  Unified Parkinson's disease Rating Scale II
UPDRS III | One month
  Unified Parkinson's disease Rating Scale III

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Frazzitta, MD, Principal Investigator — Ospedale generale di Zona "Moriggia-Pelascini", Gravedona ed Uniti 22015 - CO, Italy
Locations (1):
- Ospedale generale di zona "Moriggia-Pelascini", Gravedona, Como, Italy